CLINICAL TRIAL: NCT07315308
Title: Preoperative Ultrasound-Guided Deep Parasternal Intercostal Plane Block Reduces Intraoperative Opioid Consumption in Adults Undergoing Cardiac Surgery Via Median Sternotomy
Brief Title: Preoperative Deep Parasternal Intercostal Plane Block and Intraoperative Opioid Use in Cardiac Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziantep City Hospital (Other)
Responsible Party: Principal Investigator, Burak Cemil Balık, Attending Anesthesiologist, Gaziantep City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 390
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain; Sternotomy; Opioid Consumption; Intraoperative Pain Control
Keywords: Deep parasternal intercostal plane block; Parasternal block; Ultrasound-guided regional anesthesia; Sternotomy analgesia; Cardiac surgery pain management; Opioid-sparing analgesia; Multimodal analgesia; Anterior chest wall block; Regional anesthesia in cardiac surgery; Intraoperative Pain; Intraoperative Opioid Consumption
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to one of two parallel groups. The intervention group will receive a preoperative bilateral ultrasound-guided deep parasternal intercostal plane block in addition to standardized multimodal analgesia, while the control group will receive standardized multimodal analgesia alone. All participants will undergo elective cardiac surgery via median sternotomy under general anesthesia. Outcomes will be assessed intraoperatively and during the first 24 hours postoperatively.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to group allocation, as the deep parasternal intercostal plane block will be performed after induction of general anesthesia. Postoperative outcome assessments, including pain scores, opioid consumption, and time to extubation, will be conducted by an independent outcome assessor who is blinded to group assignment. The anesthesiologist performing the regional block will not be blinded due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep Parasternal Intercostal Plane Block Group (Experimental): Participants in this arm will receive a bilateral ultrasound-guided deep parasternal intercostal plane block following induction of general anesthesia, in addition to standard multimodal perioperative analgesia. The block will be performed in the parasternal region under real-time ultrasound guidance by injection of local anesthetic into the fascial plane between the internal intercostal and transversus thoracis muscles.
  Interventions: Procedure: Deep Parasternal Intercostal Plane Block
- Standard Analgesia (Control) Group (Active Comparator): Participants in this arm will receive standard multimodal perioperative analgesia according to institutional cardiac anesthesia protocols. No regional anesthesia techniques, including parasternal plane blocks, will be performed.
  Interventions: Procedure: Deep Parasternal Intercostal Plane Block; Other: Standard Multimodal Analgesia

INTERVENTIONS:
Procedure: Deep Parasternal Intercostal Plane Block — Bilateral ultrasound-guided deep parasternal intercostal plane block performed after induction of general anesthesia, with injection of local anesthetic into the fascial plane between the internal intercostal and transversus thoracis muscles for postoperative analgesia.
Other: Standard Multimodal Analgesia — Standard postoperative multimodal analgesia administered according to institutional cardiac anesthesia protocols, without any regional anesthesia technique.
  Arms: Standard Analgesia (Control) Group

SUMMARY:
Median sternotomy is commonly used in cardiac surgery and is associated with significant intraoperative and postoperative pain, often requiring substantial opioid administration. High opioid use during cardiac surgery may contribute to adverse effects such as respiratory depression, delayed extubation, postoperative nausea and vomiting, and prolonged intensive care unit stay. Therefore, effective opioid-sparing strategies are an important component of modern perioperative care.

The deep parasternal intercostal plane (DPIP) block is a regional anesthesia technique that targets the anterior cutaneous branches of the intercostal nerves, which are responsible for transmitting pain from the sternum and adjacent tissues. When performed under ultrasound guidance, this block allows precise local anesthetic deposition while minimizing the risk of pleural or vascular injury.

The purpose of this randomized controlled study is to evaluate whether a preoperative ultrasound-guided DPIP block reduces intraoperative opioid consumption in adult patients undergoing elective cardiac surgery via median sternotomy. Patients will be randomly assigned to receive either a bilateral DPIP block in addition to standard general anesthesia or standard general anesthesia alone.

The primary outcome of the study is total intraoperative opioid consumption. Secondary outcomes include time to extubation, postoperative opioid consumption within the first 24 hours, postoperative pain scores, and the incidence of opioid-related adverse effects. The results of this study may help define the role of the DPIP block as part of a multimodal, opioid-sparing analgesic strategy in cardiac surgery.

DETAILED DESCRIPTION:
Adequate pain control during and after cardiac surgery via median sternotomy remains challenging despite advances in perioperative care. Opioids continue to be the mainstay of analgesia; however, excessive intraoperative opioid administration has been associated with delayed extubation, respiratory complications, postoperative nausea and vomiting, and prolonged intensive care unit stay. As part of enhanced recovery protocols, regional anesthesia techniques that provide effective opioid-sparing analgesia are increasingly emphasized.

The deep parasternal intercostal plane (DPIP) block is a relatively novel ultrasound-guided regional anesthesia technique that targets the anterior cutaneous branches of the intercostal nerves within the fascial plane between the internal intercostal and transversus thoracis muscles. Compared with more proximal neuraxial or paravertebral techniques, the DPIP block offers a more localized and anatomically specific approach to sternotomy-related pain while potentially reducing the risk of serious complications.

In this prospective, randomized controlled trial, adult patients scheduled for elective cardiac surgery via median sternotomy will be allocated to one of two parallel groups. Patients in the intervention group will receive a bilateral ultrasound-guided DPIP block performed preoperatively after induction of general anesthesia, in addition to standardized general anesthesia management. Patients in the control group will receive standardized general anesthesia alone, without a regional block. Perioperative anesthetic management, including opioid administration, will follow institutional protocols and will be guided by routine clinical parameters.

The primary objective of the study is to assess the effect of the preoperative DPIP block on total intraoperative opioid consumption. Secondary objectives include evaluation of early recovery parameters such as time to extubation, postoperative opioid requirements within the first 24 hours, postoperative pain intensity, and the occurrence of opioid-related adverse events. Safety outcomes related to the block procedure will also be recorded.

This study is designed to provide clinically relevant data on the role of the DPIP block as part of a multimodal analgesic strategy in cardiac surgery. By focusing on intraoperative opioid consumption and early recovery outcomes, the trial aims to clarify whether preoperative application of this targeted regional technique can contribute to improved perioperative management and opioid-sparing anesthesia in patients undergoing median sternotomy.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 to 65 years Scheduled to undergo elective cardiac surgery via median sternotomy Planned general anesthesia Able to provide written informed consent

Exclusion Criteria:

Known allergy or contraindication to local anesthetics Coagulation disorders or ongoing anticoagulant therapy that contraindicates regional anesthesia Infection at or near the planned injection site Pre-existing chronic pain conditions requiring long-term opioid use Severe cognitive impairment or inability to communicate pain intensity Emergency surgery Refusal or inability to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Total Intraoperative Opioid Consumption | From induction of general anesthesia until completion of surgery
  Total amount of opioids administered intraoperatively, expressed as intravenous fentanyl equivalents (µg), adjusted for body weight (µg/kg), recorded from anesthesia records.

SECONDARY OUTCOMES:
Intraoperative Hemodynamic Stability | During surgery
  Incidence of intraoperative hemodynamic instability, defined as the need for additional opioid administration or vasoactive support in response to surgical stimulation, recorded from anesthesia records.
Time to Extubation | From completion of surgery to successful tracheal extubation in the intensive care unit
  Time elapsed between the end of surgery and successful tracheal extubation, recorded in minutes.
Postoperative Opioid Consumption | First 24 hours postoperatively
  Cumulative amount of opioids administered during the first 24 postoperative hours, expressed as intravenous morphine equivalents (mg), obtained from medical records.
Time to First Rescue Analgesia | Up to 24 hours postoperatively
  Time elapsed from arrival in the intensive care unit to the administration of the first rescue analgesic medication.
Block-Related Complications | Intraoperative period and first 24 postoperative hours
  Incidence of complications related to the parasternal intercostal plane block, including but not limited to pneumothorax, vascular puncture, local anesthetic systemic toxicity, and infection.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared, as the study is a single-center clinical trial and data sharing was not included in the original study protocol or approved by the institutional ethics committee. De-identified aggregate data will be reported in scientific publications.

REFERENCES:
- [Background] Medeiros HJS, Rodrigue ACLF, Mueller A, Korn E, Sabouri AS. Analgesic efficacy of parasternal intercostal plane block for midline sternotomy in adult cardiac surgery: A systematic review and meta-analysis of randomized controlled trials. J Biol Methods. 2024 Nov 14;12(1):e99010033. doi: 10.14440/jbm.2024.0070. eCollection 2025. PMID 40200942
- [Background] Wong HMK, Chen PY, Tang GCC, Chiu SLC, Mok LYH, Au SSW, Wong RHL. Deep Parasternal Intercostal Plane Block for Intraoperative Pain Control in Cardiac Surgical Patients for Sternotomy: A Prospective Randomized Controlled Trial. J Cardiothorac Vasc Anesth. 2024 Mar;38(3):683-690. doi: 10.1053/j.jvca.2023.11.038. Epub 2023 Nov 30. PMID 38148266
- [Background] Li Q, Liao Y, Wang X, Zhan M, Xiao L, Chen Y. Efficacy of bilateral catheter superficial parasternal intercostal plane blocks using programmed intermittent bolus for opioid-sparing postoperative analgesia in cardiac surgery with sternotomy: A randomized, double-blind, placebo-controlled trial. J Clin Anesth. 2024 Aug;95:111430. doi: 10.1016/j.jclinane.2024.111430. Epub 2024 Mar 26. PMID 38537393